CLINICAL TRIAL: NCT03869268
Title: The Impact of Aspirin Dose Modification on the Innate Immune Response - Will Lower Dose Aspirin Therapy Reduce the Response to Endotoxin
Acronym: WILLOW TREE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH20370
Record Dates: First submitted 2018-12-04; First posted 2019-03-11 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Intervention Model Description: This trial is a randomised controlled hybrid parallel-group and crossover study.
Masking Description: Masking is not applicable for this trial as this is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- No Drug (Active Comparator): Patients will be randomised to receive no drug for the first medication period (10 days).
  Patient will then be allocated to receive ticagrelor 90mg twice daily for the second medication period (10 days)
  Interventions: Drug: Ticagrelor
- Ticagrelor 180 mg (Active Comparator): Participants will be randomised to receive loading dose of ticagrelor 180 mg on the last day of the first medication period (10-14 days).
  Participants will then be allocated to receive no aspirin but a loading dose of ticagrelor 180 mg on the last day of treatment for the second medication period (10-14 days).
  Interventions: Drug: Ticagrelor
- Aspirin 20mg (Active Comparator): Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10 days).
  Participants will then be allocated to receive aspirin 20 mg twice daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 20 mg & Ticagrelor 180 mg (Active Comparator): Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10-14 days).
  Participants will then be allocated to receive aspirin 20 mg twice daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 75 mg (Active Comparator): Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days).
  Participants will then be allocated to receive aspirin 75 mg once daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 75 mg & Ticagrelor 180 mg (Active Comparator): Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Participants will then be allocated to receive aspirin 75 mg once daily for the second medication period (10-14 days).
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 300 mg (Active Comparator): Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10 days).
  Participants will then be allocated to receive aspirin 300 mg once daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 300 mg & Ticagrelor 180 mg (Active Comparator): Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10-14 days) plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Participants will then be allocated to receive aspirin 300 mg once daily for the second medicaion period (10-14 days).
  Interventions: Drug: Aspirin; Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin — Aspirin will be allocated in different doses and will be used in conjunction with ticagrelor depending on the arm of the trial the participant is randomised to. The different doses are as follows: 20 mg, 75 mg and 300 mg.
  Arms: Aspirin 20 mg & Ticagrelor 180 mg; Aspirin 20mg; Aspirin 300 mg; Aspirin 300 mg & Ticagrelor 180 mg; Aspirin 75 mg; Aspirin 75 mg & Ticagrelor 180 mg
Drug: Ticagrelor — Ticagrelor will be allocated as a single loading dose of 180 mg (2 x 90 mg orodispersible tablets) and will be used in conjunction with aspirin depending on the arm of the trial the participant is randomised to.

SUMMARY:
Heart attacks are usually caused by clots in a coronary artery, depriving the heart muscle of blood. Platelets are the main type of blood cell causing clots to form and physicians typically give a combination of two anti-platelet drugs, aspirin and ticagrelor, to treat this. However, aspirin and ticagrelor have effects not just on the platelets but also on the immune system. The investigator has been investigating the effects of different doses of aspirin in heart attack participants when taken alongside ticagrelor, and have found that a new, lower dose of aspirin given twice daily, rather than the usual standard dose once daily, reduces the tendency to bleed whilst on treatment. The investigators are hoping to study the wider effects of different aspirin doses, with and without ticagrelor, and have therefore developed this study.

During the two periods of the study, the investigator will give healthy volunteers a combinations of these medications and then stimulate their immune system, in order to see if the medications affect the immune response. The study will involve a period of medication for 10-14 days followed by a day in hospital stimulating the immune system with an injection into the bloodstream of a substance known as endotoxin, which causes temporary flu-like symptoms, followed by blood and urine tests. The investigator will then repeat the process, after a minimum of five weeks, taking a different medication combination and having a further endotoxin injection. The investigator will also keep in contact by telephone until 2 weeks after the end of the medication to ensure participant remain well.

DETAILED DESCRIPTION:
Potential participants will contact the research team in response to advertisement. the research team will then set up a screening appointment in the Clinical Research Facility (CRF) at the Northern general Hospital. They will be offered the chance to be sent a copy of the Participant information sheet for the study before the screening appointment, otherwise they will receive on arrival to the CRF and will be given as much time as they would like to read this.

At the screening appointment (visit 1), a medically qualified member of the research team will discuss with the potential participant the background, rationale, design, requirements and risk of the study. The potential participant will have chance to ask any questions they wish and their understanding of the key points will be checked. If they are then happy to sign the consent form, they will do so and the medically-qualified members of the research team taking consent will also sign this. The participant will receive a copy of the signed form for their records. Once written consent has been obtained, participants will be interviewed to obtain information about their demographic details, medical history and medications. They will undergo a physical examination, have their vital signs and height/weight recorded, and have blood drawn from a vein for safety tests.

At visit 2, which should occur within 14 days of visit 1 but not before the results of the safety blood tests are known, ongoing consent, any new adverse events and medication changes will be recorded. Vital signs will be checked and physical examination performed. The research team will review the results of the safety blood tests and, in combination with information collected at visit 1, determine if the participant meets all the inclusion criteria and none of the exclusion criteria, and therefore whether they can proceed to randomisation, which will be performed using an electronic (online) system designed for this purpose, sealedenvelope.com.

Participants will be randomised to receive one of the following 8 treatment regimens, for 10 days, during the first period of the study:

* no drug
* Ticagrelor 180 milligrams (mg) as a loading dose on the last day
* Aspirin 20 mg BD
* Aspirin 20 mg BD, plus ticagrelor 180 mg as a loading dose on the last day
* Aspirin 75 mg once-daily (OD)
* Aspirin 75 mg, plus ticagrelor 180 mg as a loading dose on the last day
* Aspirin 300 mg OD
* Aspirin 300 mg OD, plus ticagrelor 180 mg as a loading dose on the last day

Participants will receive the supply of study medication for the first period and will be instructed when to take this. Aspirin will be supplied as a soluble powder preparation in 100 mg sachets that will be used to prepare 20 mg, 75 mg and 300 mg doses. If required by the study to take aspirin, they will be trained in preparing the correct dose, provided with written illustrated instructions and appropriate equipment for this. They will have blood drawn and urine collected for baseline tests, and will undergo measurements of the bleeding time, whereby an inflatable cuff (of the type used for measuring blood pressure) is inflated to a low pressure around the arm, 3 small cuts in the skin of the forearm are made using sprung lancets designed to minimise discomfort, and the time taken for the cuts to stop bleeding is measured.

Participants will then take their allocated study treatment for 10-14 days (medication period 1), and will be asked not to take this on the morning of visit 3.

At visit 3, which occur after 10-14 days of study medication, participants will once again attend the CRF, this time for a full day. Ongoing consent, any new relevant adverse events and medication changes will be recorded. Participants will undergo physical examination and check of vital signs to ensure they remain well. An intravenous cannula (of the kind typically used for a 'drip') will be inserted into a vein in each arm. One cannula (cannula A) will be used for blood sampling and the other (cannula B) for injection/infusion throughout the course of the day. Blood will be drawn from cannula A for study tests, bleeding time will be measured and urine collected. Participants will then be asked to take the last dose of study medication for period 1, including, where specified by the protocol, a loading dose of ticagrelor administered in the form of 2 x 90 mg orodispersible tablets. Unused medication will be collected, counted and returned to the Northern General Pharmacy.

30 minutes later, an infusion ('drip') of normal saline will be started through cannula B to ensure participants are well hydrated. This will continue for 3 hours and 30 minutes in total. 30 minutes into the infusion, vital signs will be checked, blood will be sampled from cannula A, bleeding time will be measured and an injection of a weight-adjusted dose of sterile bacterial endotoxin will be given through cannula B.

Further blood for study tests will be drawn 0.5, 1, 1.5, 2, 3, 4 and 6 hours after the endotoxin injection. Urine will be collected 1, 2, 4 and 6 hours after the endotoxin injection, Bleeding time will be measured 3 hours after the endotoxin injection. From the time of endotoxin administration until 6 hours after it, participants will be connected to a continuous cardiac monitor, and vital signs will be checked at 0.5, 1, 1.5, 2, 3, 4 and 6 hours after the endotoxin injection. Any reportable adverse events will be recorded throughout the day. At the end of the day (6 hours after endotoxin injection) if feeling well participants will be allowed home, but if there are any concerns arrangements will be made for them to stay later, if necessary overnight, within the CRF or a ward of the Northern General Hospital.

The day after visit 3, participants will be contacted by telephone by a member of the research team (visit 4). Ongoing consent, any new relevant adverse events and medication changes will be recorded. If there are any concerns raised by the participant or investigator arrangements will be made for an in-person review by a medically qualified member of the research team in the CRF.

There will then be a break in study medication of at least five weeks. This is to ensure that any effects of the endotoxin and/or study medication have completely worn off before the next stage of the trial. At 10-14 days after visit 3, participants will be contacted by telephone by a member of the research team (visit 4). Ongoing consent, any new relevant adverse events and medication changes will be recorded. If there are any concerns raised by the participant or investigator arrangements will be made for an in-person review by a medically qualified member of the research team in the CRF.

At visit 6, participants will attend for a clinic visit in the CRF. Ongoing consent, new relevant events and medications changes will be recorded. Vital signs will be checked, physical examination performed and safety blood tests taken. A new set of medication will be provided to the participant, with appropriate training in aspirin dosing if needed. The medication that the participant will be asked to take for the next 10-14 days (medication period 2) will be determined by what they were allocated in medication period 1:

* If received no drug in period 1, to receive no aspirin in period 2 but receive a loading dose of 180 mg ticagrelor on the last day of period 2
* If received no aspirin but received a loading dose of 180 mg ticagrelor on the last day of period 1, to receive no drug in period 2
* If received aspirin 20 mg BD but no ticagrelor in period 1, to receive aspirin 20mg BD in period 2 plus a loading dose of 180 mg ticagrelor on the last day of period 2
* If received aspirin 20 mg BD plus a loading dose of 180 mg ticagrelor on the last day of period 1, to receive aspirin 20 mg BD and no ticagrelor in period 2.
* If received aspirin 75 mg OD but no ticagrelor in period 1, to receive aspirin 75 mg OD in period 2 plus a loading dose of 180 mg ticagrelor on the last day of period 2
* If received aspirin 75 mg OD plus a loading dose of 180 mg ticagrelor on the last day of period 1, to receive aspirin 75 mg OD and no ticagrelor in period 2.
* If received aspirin 300 mg OD but no ticagrelor in period 1, to receive aspirin 300 mg OD in period 2 plus a loading dose of 180 mg ticagrelor on the last day of period 2
* If received aspirin 300 mg OD plus a loading dose of 180 mg ticagrelor on the last day of period 1, to receive aspirin 300 mg OD and no ticagrelor in period 2.

Participants will then take their allocated study treatment for 10-14 days (medication period 2) and will be asked not to take this on the morning of visit 7.

Visits 7, 8 and 9 will be another full day visit to the CRF followed by a telephone call the next day and after 10-14 days. These will follow exactly the same process as visit 3, 4 and 5. At this point their involvement in the study will end and they will be thanked for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, or female subjects not of childbearing potential (either surgically sterile or post-menopausal)]
* Age between 18 and 65 years inclusive
* Non-smokers
* Body mass index (BMI) between 18 and 28 kg/m2 inclusive, with a body weight between 60-100 kg
* In good health as determined by a medical history, physical examination, vital signs and clinical laboratory test results, including renal and liver function, and full blood count
* Provision of informed consent before any trial-related activity

Exclusion Criteria:

* Any history of cancer, diabetes or, in the opinion of the investigator, clinically-significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, haematological, dermatological, neurological, psychiatric or other major disorders
* Any history of either significant multiple drug allergies or known allergy to the study drugs or any medicine chemically related to the study drugs
* A clinically-significant illness within 4 weeks of randomisation
* Any clinically-significant abnormal laboratory test results at screening in the opinion of the investigator
* A supine blood pressure at screening, after resting for 5 minutes, higher than 150/90 mmHg or lower than 105/65 mmHg
* A supine heart rate at screening, after resting for 5 minutes, outside the range of 50-100 beats/min
* Receipt of any prescribed or over-the-counter systemic or topical medication within 48 hours prior to the start of dosing
* Planned or expected requirement, during the next 3 months (at randomisation, or 3 weeks at the start of period 2), for any systemic or topical prescribed drug, or for systemic or topical over-the-counter NSAID, corticosteroid, anthihistamine or any other drug that could affect inflammation, thrombosis or haemostasis in the opinion of the investigator.
* Receipt of an investigational medicinal product within the previous four months (new chemical entity) or three months (licensed product) or subjects who have received a vaccine within three weeks preceding the start of dosing. When reconfirming eligibility at the start of period 2, receipt of aspirin, ticagrelor or endotoxin during period 1 of this study will not be counted for this purpose.
* Any donation of blood or plasma in the month preceding the start of dosing.
* A history of alcohol or drug abuse
* Mental incapacity or language barriers that preclude adequate understanding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Jackson SP. Arterial thrombosis--insidious, unpredictable and deadly. Nat Med. 2011 Nov 7;17(11):1423-36. doi: 10.1038/nm.2515. PMID 22064432
- [Background] Luc G, Bard JM, Juhan-Vague I, Ferrieres J, Evans A, Amouyel P, Arveiler D, Fruchart JC, Ducimetiere P; PRIME Study Group. C-reactive protein, interleukin-6, and fibrinogen as predictors of coronary heart disease: the PRIME Study. Arterioscler Thromb Vasc Biol. 2003 Jul 1;23(7):1255-61. doi: 10.1161/01.ATV.0000079512.66448.1D. Epub 2003 May 29. PMID 12775578
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Solari HP, Ventura MP, Orellana ME, Novais GA, Cheema DP, Burnier MN Jr. Histopathological study of lesions of the caruncle: a 15-year single center review. Diagn Pathol. 2009 Aug 31;4:29. doi: 10.1186/1746-1596-4-29. PMID 19719846
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Thomas MR, Outteridge SN, Ajjan RA, Phoenix F, Sangha GK, Faulkner RE, Ecob R, Judge HM, Khan H, West LE, Dockrell DH, Sabroe I, Storey RF. Platelet P2Y12 Inhibitors Reduce Systemic Inflammation and Its Prothrombotic Effects in an Experimental Human Model. Arterioscler Thromb Vasc Biol. 2015 Dec;35(12):2562-70. doi: 10.1161/ATVBAHA.115.306528. Epub 2015 Oct 29. PMID 26515417
- [Background] Patrono C, Morais J, Baigent C, Collet JP, Fitzgerald D, Halvorsen S, Rocca B, Siegbahn A, Storey RF, Vilahur G. Antiplatelet Agents for the Treatment and Prevention of Coronary Atherothrombosis. J Am Coll Cardiol. 2017 Oct 3;70(14):1760-1776. doi: 10.1016/j.jacc.2017.08.037. PMID 28958334
- [Background] Patrono C. Aspirin as an antiplatelet drug. N Engl J Med. 1994 May 5;330(18):1287-94. doi: 10.1056/NEJM199405053301808. No abstract available. PMID 8145785
- [Background] Randomised trial of intravenous streptokinase, oral aspirin, both, or neither among 17,187 cases of suspected acute myocardial infarction: ISIS-2. ISIS-2 (Second International Study of Infarct Survival) Collaborative Group. Lancet. 1988 Aug 13;2(8607):349-60. PMID 2899772
- [Background] Belch J, MacCuish A, Campbell I, Cobbe S, Taylor R, Prescott R, Lee R, Bancroft J, MacEwan S, Shepherd J, Macfarlane P, Morris A, Jung R, Kelly C, Connacher A, Peden N, Jamieson A, Matthews D, Leese G, McKnight J, O'Brien I, Semple C, Petrie J, Gordon D, Pringle S, MacWalter R; Prevention of Progression of Arterial Disease and Diabetes Study Group; Diabetes Registry Group; Royal College of Physicians Edinburgh. The prevention of progression of arterial disease and diabetes (POPADAD) trial: factorial randomised placebo controlled trial of aspirin and antioxidants in patients with diabetes and asymptomatic peripheral arterial disease. BMJ. 2008 Oct 16;337:a1840. doi: 10.1136/bmj.a1840. PMID 18927173
- [Background] Pignone M, Alberts MJ, Colwell JA, Cushman M, Inzucchi SE, Mukherjee D, Rosenson RS, Williams CD, Wilson PW, Kirkman MS. Aspirin for primary prevention of cardiovascular events in people with diabetes: a position statement of the American Diabetes Association, a scientific statement of the American Heart Association, and an expert consensus document of the American College of Cardiology Foundation. Circulation. 2010 Jun 22;121(24):2694-701. doi: 10.1161/CIR.0b013e3181e3b133. Epub 2010 May 27. No abstract available. PMID 20508178
- [Background] Ogawa H, Nakayama M, Morimoto T, Uemura S, Kanauchi M, Doi N, Jinnouchi H, Sugiyama S, Saito Y; Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes (JPAD) Trial Investigators. Low-dose aspirin for primary prevention of atherosclerotic events in patients with type 2 diabetes: a randomized controlled trial. JAMA. 2008 Nov 12;300(18):2134-41. doi: 10.1001/jama.2008.623. Epub 2008 Nov 9. PMID 18997198
- [Background] Ikeda Y, Shimada K, Teramoto T, Uchiyama S, Yamazaki T, Oikawa S, Sugawara M, Ando K, Murata M, Yokoyama K, Ishizuka N. Low-dose aspirin for primary prevention of cardiovascular events in Japanese patients 60 years or older with atherosclerotic risk factors: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2510-20. doi: 10.1001/jama.2014.15690. PMID 25401325
- [Background] Gaziano JM, Brotons C, Coppolecchia R, Cricelli C, Darius H, Gorelick PB, Howard G, Pearson TA, Rothwell PM, Ruilope LM, Tendera M, Tognoni G; ARRIVE Executive Committee. Use of aspirin to reduce risk of initial vascular events in patients at moderate risk of cardiovascular disease (ARRIVE): a randomised, double-blind, placebo-controlled trial. Lancet. 2018 Sep 22;392(10152):1036-1046. doi: 10.1016/S0140-6736(18)31924-X. Epub 2018 Aug 26. PMID 30158069
- [Background] Paul-Clark MJ, Van Cao T, Moradi-Bidhendi N, Cooper D, Gilroy DW. 15-epi-lipoxin A4-mediated induction of nitric oxide explains how aspirin inhibits acute inflammation. J Exp Med. 2004 Jul 5;200(1):69-78. doi: 10.1084/jem.20040566. PMID 15238606
- [Background] Kiers D, van der Heijden WA, van Ede L, Gerretsen J, de Mast Q, van der Ven AJ, El Messaoudi S, Rongen GA, Gomes M, Kox M, Pickkers P, Riksen NP. A randomised trial on the effect of anti-platelet therapy on the systemic inflammatory response in human endotoxaemia. Thromb Haemost. 2017 Aug 30;117(9):1798-1807. doi: 10.1160/TH16-10-0799. Epub 2017 Jul 6. PMID 28692111
- [Background] McAdam BF, Mardini IA, Habib A, Burke A, Lawson JA, Kapoor S, FitzGerald GA. Effect of regulated expression of human cyclooxygenase isoforms on eicosanoid and isoeicosanoid production in inflammation. J Clin Invest. 2000 May;105(10):1473-82. doi: 10.1172/JCI9523. PMID 10811855
- [Background] Birrell MA, Maher SA, Dekkak B, Jones V, Wong S, Brook P, Belvisi MG. Anti-inflammatory effects of PGE2 in the lung: role of the EP4 receptor subtype. Thorax. 2015 Aug;70(8):740-7. doi: 10.1136/thoraxjnl-2014-206592. Epub 2015 May 4. PMID 25939749
- [Background] Na YR, Jung D, Yoon BR, Lee WW, Seok SH. Endogenous prostaglandin E2 potentiates anti-inflammatory phenotype of macrophage through the CREB-C/EBP-beta cascade. Eur J Immunol. 2015 Sep;45(9):2661-71. doi: 10.1002/eji.201545471. Epub 2015 Jul 20. PMID 26118414
- [Background] Chow JC, Young DW, Golenbock DT, Christ WJ, Gusovsky F. Toll-like receptor-4 mediates lipopolysaccharide-induced signal transduction. J Biol Chem. 1999 Apr 16;274(16):10689-92. doi: 10.1074/jbc.274.16.10689. PMID 10196138
- [Background] Brasier AR. The nuclear factor-kappaB-interleukin-6 signalling pathway mediating vascular inflammation. Cardiovasc Res. 2010 May 1;86(2):211-8. doi: 10.1093/cvr/cvq076. Epub 2010 Mar 3. PMID 20202975
- [Background] Degraaf AJ, Zaslona Z, Bourdonnay E, Peters-Golden M. Prostaglandin E2 reduces Toll-like receptor 4 expression in alveolar macrophages by inhibition of translation. Am J Respir Cell Mol Biol. 2014 Aug;51(2):242-50. doi: 10.1165/rcmb.2013-0495OC. PMID 24601788
- [Background] Lee KM, Seong SY. Partial role of TLR4 as a receptor responding to damage-associated molecular pattern. Immunol Lett. 2009 Jun 30;125(1):31-9. doi: 10.1016/j.imlet.2009.05.006. Epub 2009 Jun 6. PMID 19501120
- [Background] Smiley ST, King JA, Hancock WW. Fibrinogen stimulates macrophage chemokine secretion through toll-like receptor 4. J Immunol. 2001 Sep 1;167(5):2887-94. doi: 10.4049/jimmunol.167.5.2887. PMID 11509636
- [Background] Smeeth L, Thomas SL, Hall AJ, Hubbard R, Farrington P, Vallance P. Risk of myocardial infarction and stroke after acute infection or vaccination. N Engl J Med. 2004 Dec 16;351(25):2611-8. doi: 10.1056/NEJMoa041747. PMID 15602021
- [Background] Morris T, Stables M, Hobbs A, de Souza P, Colville-Nash P, Warner T, Newson J, Bellingan G, Gilroy DW. Effects of low-dose aspirin on acute inflammatory responses in humans. J Immunol. 2009 Aug 1;183(3):2089-96. doi: 10.4049/jimmunol.0900477. Epub 2009 Jul 13. PMID 19597002
- [Background] Layne K, Di Giosia P, Ferro A, Passacquale G. Anti-platelet drugs attenuate the expansion of circulating CD14highCD16+ monocytes under pro-inflammatory conditions. Cardiovasc Res. 2016 Jul 1;111(1):26-33. doi: 10.1093/cvr/cvw089. Epub 2016 Apr 26. PMID 27118470
- [Background] Serezani CH, Lewis C, Jancar S, Peters-Golden M. Leukotriene B4 amplifies NF-kappaB activation in mouse macrophages by reducing SOCS1 inhibition of MyD88 expression. J Clin Invest. 2011 Feb;121(2):671-82. doi: 10.1172/JCI43302. Epub 2011 Jan 4. PMID 21206089
- [Background] Vranckx P, Valgimigli M, Juni P, Hamm C, Steg PG, Heg D, van Es GA, McFadden EP, Onuma Y, van Meijeren C, Chichareon P, Benit E, Mollmann H, Janssens L, Ferrario M, Moschovitis A, Zurakowski A, Dominici M, Van Geuns RJ, Huber K, Slagboom T, Serruys PW, Windecker S; GLOBAL LEADERS Investigators. Ticagrelor plus aspirin for 1 month, followed by ticagrelor monotherapy for 23 months vs aspirin plus clopidogrel or ticagrelor for 12 months, followed by aspirin monotherapy for 12 months after implantation of a drug-eluting stent: a multicentre, open-label, randomised superiority trial. Lancet. 2018 Sep 15;392(10151):940-949. doi: 10.1016/S0140-6736(18)31858-0. Epub 2018 Aug 27. PMID 30166073
- [Background] Baber U, Dangas G, Cohen DJ, Gibson CM, Mehta SR, Angiolillo DJ, Pocock SJ, Krucoff MW, Kastrati A, Ohman EM, Steg PG, Badimon J, Zafar MU, Chandrasekhar J, Sartori S, Aquino M, Mehran R. Ticagrelor with aspirin or alone in high-risk patients after coronary intervention: Rationale and design of the TWILIGHT study. Am Heart J. 2016 Dec;182:125-134. doi: 10.1016/j.ahj.2016.09.006. Epub 2016 Sep 28. PMID 27914492
- [Background] Teng R, Maya J, Butler K. Evaluation of the pharmacokinetics and pharmacodynamics of ticagrelor co-administered with aspirin in healthy volunteers. Platelets. 2013;24(8):615-24. doi: 10.3109/09537104.2012.748185. Epub 2012 Dec 18. PMID 23249161
- [Background] Scavone M, Femia EA, Caroppo V, Cattaneo M. Inhibition of the platelet P2Y12 receptor for adenosine diphosphate does not impair the capacity of platelet to synthesize thromboxane A2. Eur Heart J. 2016 Nov 21;37(44):3347-3356. doi: 10.1093/eurheartj/ehv551. Epub 2015 Oct 29. PMID 26516174
- [Background] Mahaffey KW, Wojdyla DM, Carroll K, Becker RC, Storey RF, Angiolillo DJ, Held C, Cannon CP, James S, Pieper KS, Horrow J, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor compared with clopidogrel by geographic region in the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2011 Aug 2;124(5):544-54. doi: 10.1161/CIRCULATIONAHA.111.047498. Epub 2011 Jun 27. PMID 21709065
- [Background] Suffredini AF, Hochstein HD, McMahon FG. Dose-related inflammatory effects of intravenous endotoxin in humans: evaluation of a new clinical lot of Escherichia coli O:113 endotoxin. J Infect Dis. 1999 May;179(5):1278-82. doi: 10.1086/314717. PMID 10191237
- [Background] Rittig N, Thomsen HH, Bach E, Jorgensen JO, Moller N. Hormone and Cytokine Responses to Repeated Endotoxin Exposures-No Evidence of Endotoxin Tolerance After 5 Weeks in Humans. Shock. 2015 Jul;44(1):32-5. doi: 10.1097/SHK.0000000000000384. PMID 25895146

RESULTS

PARTICIPANT FLOW:
Groups:
- No Drug, no Drug Plus Loading Dose Ticagrelor 180 mg: Patients will be randomised to receive no drug for the first medication period (10 days).
  Patient will then be allocated to receive no drug for the second medication period (10 days) and Ticagrelor will be allocated as a single loading dose of 180 mg (2 x 90 mg orodispersible tablets) on the second endotoxin visit.
- No Drug Plus Loading Dose Ticagrelor 180mg, no Drug: Participants will be randomised to receive loading dose of ticagrelor 180 mg on the last day of the first medication period (10-14 days).
  Participants will then be allocated to receive no aspirin and no ticagrelor loading dose for the second medication period (10-14 days).
- Aspirin 20mg BD, Then Aspirin 20mg BD Plus Loading Dose Ticagrelor 180mg: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10 days).
  Participants will then be allocated to receive aspirin 20 mg twice daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
- Aspirin 20mg BD & Loading Dose Ticagrelor 180mg, Then Aspirin 20mg BD no Loading Dose: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10-14 days)plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Participants will then be allocated to receive aspirin 20 mg twice daily for the second medication period (10-14 days), with no loading dose on endotoxin challenge day.
- Aspirin 75mg OD no Loading Dose of Ticagrelor, Then Aspirin 75mg & Loading Dose Ticagrelor 180mg: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days).
  Participants will then be allocated to receive aspirin 75 mg once daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
- Aspirin 75mg OD & Loading Dose Ticagrelor 180mg, Then Aspirin 75mg, no Loading Dose of Ticagrelor: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days),with a loading dose of ticagrelor 180 mg on the last day of the period.
  Participants will then be allocated to receive aspirin 75 mg once daily for the second medication period (10-14 days), no loading dose of ticagrelor.
- Aspirin 300mg OD, Then Aspirin 300mg OD Plus Loading Dose Ticagrelor 180mg: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10 days).
  Participants will then be allocated to receive aspirin 300 mg once daily for the second medication period (10-14 days), plus a loading dose of ticagrelor 180 mg on the last day of the period.
- Aspirin 300mg & Ticagrelor 180mg Loading Dose, Then Aspirin 300mg OD no Loading Dose Ticagrelor: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10-14 days) plus a loading dose of ticagrelor 180 mg on the last day of the period.
  Participants will then be allocated to receive aspirin 300 mg once daily for the second medicaion period (10-14 days).
Period: Intervention + Endotoxin
Arm/Group | No Drug, no Drug Plus Loading Dose Ticagrelor 180 mg | No Drug Plus Loading Dose Ticagrelor 180mg, no Drug | Aspirin 20mg BD, Then Aspirin 20mg BD Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg, Then Aspirin 20mg BD no Loading Dose | Aspirin 75mg OD no Loading Dose of Ticagrelor, Then Aspirin 75mg & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg, Then Aspirin 75mg, no Loading Dose of Ticagrelor | Aspirin 300mg OD, Then Aspirin 300mg OD Plus Loading Dose Ticagrelor 180mg | Aspirin 300mg & Ticagrelor 180mg Loading Dose, Then Aspirin 300mg OD no Loading Dose Ticagrelor
Started | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Completed | 8 | 9 | 9 | 9 | 8 | 8 | 9 | 7
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Period: Intervention + Endotoxin (Post Washout)
Arm/Group | No Drug, no Drug Plus Loading Dose Ticagrelor 180 mg | No Drug Plus Loading Dose Ticagrelor 180mg, no Drug | Aspirin 20mg BD, Then Aspirin 20mg BD Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg, Then Aspirin 20mg BD no Loading Dose | Aspirin 75mg OD no Loading Dose of Ticagrelor, Then Aspirin 75mg & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg, Then Aspirin 75mg, no Loading Dose of Ticagrelor | Aspirin 300mg OD, Then Aspirin 300mg OD Plus Loading Dose Ticagrelor 180mg | Aspirin 300mg & Ticagrelor 180mg Loading Dose, Then Aspirin 300mg OD no Loading Dose Ticagrelor
Started | 7 | 9 | 8 | 8 | 5 | 8 | 8 | 7
Completed | 7 | 9 | 8 | 8 | 5 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Drug, no Drug Plus Loading Dose Ticagrelor 180 mg | No Drug Plus Loading Dose Ticagrelor 180mg, no Drug | Aspirin 20mg BD, Then Aspirin 20mg BD Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg, Then Aspirin 20mg BD no Loading Dose | Aspirin 75mg OD no Loading Dose of Ticagrelor, Then Aspirin 75mg & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg, Then Aspirin 75mg, no Loading Dose of Ticagrelor | Aspirin 300mg OD, Then Aspirin 300mg OD Plus Loading Dose Ticagrelor 180mg | Aspirin 300mg & Ticagrelor 180mg Loading Dose, Then Aspirin 300mg OD no Loading Dose Ticagrelor | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 6
  Male | 9 | 8 | 9 | 8 | 6 | 9 | 9 | 8 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 7 | 9 | 7 | 8 | 7 | 7 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Assess Inflammatory Response to Intravenous Endotoxin
Description: plasma TNF-α at 2 hours post-injection of 2 ng/kg endotoxin compared between participants receiving no IMP, aspirin (Aspirin lysine) 20 mg BD, aspirin (Aspirin lysine) 75 mg OD and aspirin (Aspirin lysine) 300 mg OD.
Time Frame: 2 hours post endotoxin injection
Population: all participants that completed one or both endotoxin challenge days
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- No Drug: Patients will be randomised to receive no drug for the first medication period (10 days) and will not receive any drug on the endotoxin challenge day
- No Drug Plus Loading Dose Ticagrelor 180mg: Participants will be randomised to receive loading dose of ticagrelor 180 mg on the last day of the first medication period (10-14 days).
- Aspirin 20mg BD: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10 days) and will not receive study drugs on the endotoxin challenge day
- Aspirin 20mg BD & Loading Dose Ticagrelor 180mg: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10-14 days)plus a loading dose of ticagrelor 180 mg on the last day of the period.
- Aspirin 75mg OD no Loading Dose of Ticagrelor: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days) and no study drug on endotoxin challenge day
- Aspirin 75mg OD & Loading Dose Ticagrelor 180mg: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days),with a loading dose of ticagrelor 180 mg on the last day of the period.
- Aspirin 300mg OD: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10 days) and no study drug on endotoxin challenge day
- Aspirin 300mg & Ticagrelor 180mg Loading Dose: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10-14 days) plus a loading dose of ticagrelor 180 mg on the last day of the period.
Arm/Group | No Drug | No Drug Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD no Loading Dose of Ticagrelor | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg | Aspirin 300mg OD | Aspirin 300mg & Ticagrelor 180mg Loading Dose
Number analyzed (Participants) | 17 | 16 | 17 | 17 | 16 | 14 | 15 | 15
pg/ml | 167.53 (186.17) | 111.05 (154.48) | 254.92 (236.79) | 128.73 (162.22) | 103.72 (141.36) | 72.95 (77.78) | 156.17 (141.28) | 126.66 (194.96)

2. Secondary Outcome: Serum CRP Changes
Description: Change in serum CRP from 0 to 6 hours after endotoxin administration
Time Frame: 0 to 6 hours after endotoxin administration
Population: all participants that completed one or both endotoxin challenge days.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | No Drug | No Drug Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD no Loading Dose of Ticagrelor | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg | Aspirin 300mg OD | Aspirin 300mg & Ticagrelor 180mg Loading Dose
Number analyzed (Participants) | 17 | 17 | 18 | 17 | 16 | 16 | 15 | 16
mg/L | 2.84 (1.54) | 3.00 (2.30) | 3.61 (2.48) | 3.11 (1.08) | 3.10 (1.40) | 2.52 (1.19) | 2.94 (2.01) | 2.60 (1.83)

3. Secondary Outcome: Leukocyte Count
Description: Leukocyte count, from 0 to 6 hours after endotoxin administration
Time Frame: 0 to 6 hours after endotoxin administration
Population: Participants who completed one or both endotoxin challenge days
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | No Drug | No Drug Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD no Loading Dose of Ticagrelor | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg | Aspirin 300mg OD | Aspirin 300mg & Ticagrelor 180mg Loading Dose
Number analyzed (Participants) | 16 | 17 | 18 | 17 | 16 | 16 | 15 | 16
10^9 cells per liter | 9.28 (2.46) | 9.32 (3.38) | 10.77 (3.63) | 11.77 (2.12) | 11.09 (2.98) | 9.99 (4.42) | 9.45 (3.83) | 8.91 (3.30)

4. Secondary Outcome: Serum TXB2
Description: Serum TXB2 from 0 to 6 hours after endotoxin administration
Time Frame: 0 to 6 hours after endotoxin administration
Population: all participants who completed one or both endotoxin challenge days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | No Drug | No Drug Plus Loading Dose Ticagrelor 180mg | Aspirin 20mg BD | Aspirin 20mg BD & Loading Dose Ticagrelor 180mg | Aspirin 75mg OD no Loading Dose of Ticagrelor | Aspirin 75mg OD & Loading Dose Ticagrelor 180mg | Aspirin 300mg OD | Aspirin 300mg & Ticagrelor 180mg Loading Dose
Number analyzed (Participants) | 16 | 15 | 17 | 17 | 17 | 14 | 15 | 15
pg/ml | 389904.00 (355874.00) | 274473.00 (212718.00) | 19334.00 (46071.00) | 3538.00 (6430.00) | 1824.00 (2466.00) | 1444.00 (1375.00) | 346.60 (495.80) | 301.00 (429.20)

ADVERSE EVENTS:
Time Frame: Adverse events and reactions will be recorded and reported from randomisation to 10 days after visit 3 (1st endotoxin injection day), and from visit 6 (start of period 2) to 10 days after visit 7 (2nd endotoxin injection day) as described in the protocol. Thus adverse events occurring in the break (wash out period) between the first and second medication periods, excepting those originating in the 10 days after endotoxin injection, will not be recorded or reported as stipulated in the protocol.
Description: Adverse events not reported as they are expected as a normal response to endotoxin:
  Abnormal body temperature, except if >39 and <34oC, unless persists at 6 hours post-endotoxin /meets the criteria of SAE; Change in pulse rate, except>140 and<45 bpm/if meets criteria for SAE; Increase/decrease in blood pressure from baseline of<40 mmHg unless an SAE; Self-limiting symptoms due to endotoxaemia at discretion of investigator, unless an SAE; Changes in leukocyte/platelet count or CRP unless SAE
Groups:
- No Drug: Patients will be randomised to receive no drug for the first medication period (10 days) followed by endotoxin challenge
- No Drug Plus Ticagrelor 180mg: Participants will be randomised to receive no drug, then a loading dose of ticagrelor 180 mg on the last day of the first medication period (10-14 days) followed by endotoxin challenge
- Aspirin 20mg BD: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10 days) followed by endotoxin challenge
- Aspirin 20mg BD & Ticagrelor 180mg: Participants will be randomised to receive aspirin 20 mg twice daily for the first medication period (10-14 days) plus a loading dose of ticagrelor 180 mg on the last day of the period followed by endotoxin challenge.
- Aspirin 75mg OD: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days).
  followed by endotoxin challenge
- Aspirin 75mg OD & Ticagrelor 180mg: Participants will be randomised to receive aspirin 75 mg once daily for the first medication period (10-14 days),with a loading dose of ticagrelor 180 mg on the last day of the period followed by endotoxin challenge
- Aspirin 300mg OD: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10 days) followed by endotoxin challenge
- Aspirin 300mg OD & Ticagrelor 180mg: Participants will be randomised to receive aspirin 300 mg once daily for the first medication period (10-14 days) plus a loading dose of ticagrelor 180 mg on the last day of the period followed by endotoxin challenge
Arm/Group | No Drug | No Drug Plus Ticagrelor 180mg | Aspirin 20mg BD | Aspirin 20mg BD & Ticagrelor 180mg | Aspirin 75mg OD | Aspirin 75mg OD & Ticagrelor 180mg | Aspirin 300mg OD | Aspirin 300mg OD & Ticagrelor 180mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17 | 0/16 | 0/14 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17 | 0/16 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/17 | 3/16 | 5/17 | 4/17 | 4/16 | 5/14 | 5/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Drug (N=17) | No Drug Plus Ticagrelor 180mg (N=16) | Aspirin 20mg BD (N=17) | Aspirin 20mg BD & Ticagrelor 180mg (N=17) | Aspirin 75mg OD (N=16) | Aspirin 75mg OD & Ticagrelor 180mg (N=14) | Aspirin 300mg OD (N=15) | Aspirin 300mg OD & Ticagrelor 180mg (N=15)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pyrexia (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
hypokalaemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pinpoint pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cold sores (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
foot injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
excess phleghm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vasovagal episode (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03869268/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03869268/SAP_001.pdf